CLINICAL TRIAL: NCT03981159
Title: Effect of Exercise Training on Biochemical and Gait/Balance Parameters in Alzheimer's Patients
Brief Title: Effect of Exercise Training in Alzheimer's Patients
Acronym: ExCiTE-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, Maamer Slimani, Principal Investigator, University of Genova
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ExCiTE-A-17-0020
Record Dates: First submitted 2019-03-03; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Physical Conditioning, Human

STUDY DESIGN:
Intervention Model Description: Non-pharmacological interventional study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (under physical training) (Experimental): Subjects belonging to this arm underwent physical training for three months, twice per week (60 minutes per session).
  Interventions: Other: Physical training
- Passive group (no physical training) (No Intervention): Subjects served as controls.

INTERVENTIONS:
Other: Physical training — Physical training for three months, twice per week (60 minutes per session).
  Arms: Active group (under physical training)

SUMMARY:
The objective of this study was to examine the effects of exercise training on physical function and biochemical markers in elderly Alzheimer's disease patients.

DETAILED DESCRIPTION:
Alzheimer's disease is a neurodegenerative disease characterized by progressive and irreversible degeneration of nerve cells. The loss of these cells leads to the continuous decline in muscle function with alterations in biochemical and haematological parameters. The objective of this study was to examine the effects of exercise training on physical function and biochemical markers in elderly Alzheimer's disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with official diagnosis of Alzheimer's disease;
* Subjects with MMSE higher than12.

Exclusion Criteria:

• Subjects with MMSE below 12 (indicating severe dementia and impairment).

Ages: 80 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Tinetti test | Approximately 10-15 minutes
  The 3-likert test assesses balance and gait abilities with an individual sitting in an armless chair, rising up, staying standing, turning 360° and then sitting back down. Gait is scored over 12 and balance is scored over 16, totalling 28 points.
Berg Balance Scale | Approximately 20 minutes
  The 14-item 5-likert (from 0 to 4) scale objectively determines a patient's balance ability during a series of predetermined tasks. Scores of each item are summed up: the total score ranges from 0 to 56. The lowest the score the lowest is the level of function, the highest the score the highest is the level of function.
6-minute walking test | 6 minutes
  This test is a sub-maximal exercise used to evaluate aerobic capacity and endurance.
Timed up and go test | Approximately 14 seconds
  The test measures abilities of a patient initially in a seated position The patient is then asked to stand up up, walk 3 meters, turn around, walk back to the chair and sit down.
"Walking While Talking" test | Approximately 1 minute
  This test is a dual-task test, consisting in walking while reciting the alphabet or alternate letters of the alphabet.
Red blood cell count | Approximately 10-15 minutes
  Assessed with routine blood/biochemical assays
White blood cell count | Approximately 10-15 minutes
  Assessed with routine blood/biochemical assays
Hemoglobin | Approximately 10-15 minutes
  Assessed with routine blood/biochemical assays
Platelet count | Approximately 10-15 minutes
  Assessed with routine blood/biochemical assays
Hematocrit | Approximately 10-15 minutes
  Assessed with routine blood/biochemical assays
Triglycerides | Approximately 10-15 minutes
  Assessed with routine blood/biochemical assays
Cholesterol | Approximately 10-15 minutes
  Assessed with routine blood/biochemical assays
Total bilirubin | Approximately 10-15 minutes
  Assessed with routine blood/biochemical assays
AST (aspartate aminotransferase) | Approximately 10-15 minutes
  Assessed with routine blood/biochemical assays
ALT (alanine aminotransferase) | Approximately 10-15 minutes
  Assessed with routine blood/biochemical assays
Blood pressure | Approximately 10-15 minutes
  Assessed with routine blood/biochemical assays
Creatinine | Approximately 10-15 minutes
  Assessed with routine blood/biochemical assays
Urea | Approximately 10-15 minutes
  Assessed with routine blood/biochemical assays
Glucose | Approximately 10-15 minutes
  Assessed with routine blood/biochemical assays
Sodium | Approximately 10-15 minutes
  Assessed with routine blood/biochemical assays
Calcium | Approximately 10-15 minutes
  Assessed with routine blood/biochemical assays
Potassium | Approximately 10-15 minutes
  Assessed with routine blood/biochemical assays

CONTACTS AND LOCATIONS:
Overall Officials: Nicola L Bragazzi, MD, PhD, MPH, Principal Investigator — Universita degli Studi di Genova
Locations (1):
- University of Genova, Genoa, Italy

IPD SHARING:
Plan to Share IPD: No